CLINICAL TRIAL: NCT00689676
Title: Expressive Language and Cognitive Early Development in Very Low Birth-Weight Preterm Toddlers
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Suelly Cecilia Olivan Limongi, University of São Paulo
Other Study IDs: 280674
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Prematurity
Keywords: expressive language; cognition; early development; very low birt weight; prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study Group: 20 very low birth weight preterm toddlers
- Control Group: 20 full-term toddlers

SUMMARY:
The aim of the present study is to describe the performance of very low birth-weight preterm toddlers regarding expressive language and cognitive development during sensorimotor and beginning of pre-operational periods, as well as to compare the performance presented by these children to that presented by their full-term peers, according to Genetic Epistemology theoretical principles.

The hypothesis of this study is that very-low birth weight preterms would present a poorer performance, concerning expressive language and cognition development,than their full-term peers.

DETAILED DESCRIPTION:
Very low birth weight preterm infants are known to have risks of cognitive and behavioral problems, including learning difficulties, attention deficits and hyperactivity, as well as neuromotor deficits. Moreover, they are reported to have a high risk of speech and language impairments up to school age, even in cases where major neurological abnormalities are excluded. Impairments have been reported both in receptive and expressive language and, more specifically, in morphosyntax and naming.

ELIGIBILITY:
Study Group:

Inclusion Criteria:

* gestational age lower than 34 weeks (according to the date of last menstrual period - DLMP);
* birth weight equal or lower than 1500g;
* exposed only to Brazilian Portuguese

Exclusion Criteria:

* presence of major malformations, genetic syndromes, severe neonatal asphyxia, hearing impairment or visual impairment.

Control Group:

Inclusion Criteria:

* gestational age higher than 38 weeks;
* adequate for gestational age;
* birth weight higher than 2500g up to 3999g
* exposed only to Brazilian Portuguese

Exclusion Criteria:

* pre, peri or post natal intercurrence

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study Group:
  Very-Low Birth weight preterm newborns (mean weight: 1073g, mean gestational age: 29 3/7w), born in the Hospital of the University of São Paulo between March 2005 and February 2006, assisted in the High Risk Newborns Follow up Ambulatory of the University's Hospital.
  Control Group:
  Full-term newborns (mean weight: 3291g, mean gestational age: 39 1/7w), followed up in the Pediatrics Ambulatory of the University's Hospital and/or being assisted in the University' Hospital Nursery School.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2006-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Performance on monthly observations carried out after the initial evaluation | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Suelly CO Limongi, PhD., Study Chair — University of Sao Paulo
Locations (1):
- University's Hospital, São Paulo, São Paulo, Brazil